CLINICAL TRIAL: NCT03866954
Title: The Safety, Tolerability, Pharmacodynamics, and Efficacy of Erythrocyte Encapsulated Thymidine Phosphorylase (EE-TP) in Patients With MNGIE
Brief Title: Trial of Erythrocyte Encapsulated Thymidine Phosphorylase In Mitochondrial Neurogastrointestinal Encephalomyopathy
Acronym: TEETPIM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change of circumstances with Commercial partner
Sponsor: St George's, University of London (Other)
Collaborators: Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018.0158; 2018-003000-39 (EudraCT Number)
Record Dates: First submitted 2019-02-04; First posted 2019-03-07 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-07

CONDITIONS: Mitochondrial Diseases; Metabolic Disease; Inborn Errors of Metabolism
Keywords: neuropathy; gastrointestinal disease; thymidine phosphorylase; enyme replacement
MeSH Terms: conditions — Mitochondrial Diseases; Metabolic Diseases; Metabolism, Inborn Errors; Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: This will be a multi-centre, multiple dose, open label study to investigate the safety, tolerability, PD, and efficacy of EE TP in patients with MNGIE. The study will be conducted in an open label manner with all patients receiving EE TP.
  The study will enrol 12 adult treatment naïve patients with MNGIE, aged 18 years or older at Screening. With IDMC approval, a further four juvenile patients (aged 16-17) will be recruited after at least 24 patient-months exposure to treatment. With IDMC approval, a further four juvenile patients (aged 12-15) will be recruited after at least 24 patient-months exposure to treatment in the 16-17 year old patient group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous administration of EE-TP (Experimental): Intravenous administration of EE-TP. The starting dose will be Dose Level 1, with potential subsequent dose levels of Dose Level 2 and Dose Level 3 dependent on whether metabolic correction is achieved or not.
  Interventions: Combination Product: EE-TP

INTERVENTIONS:
Combination Product: EE-TP — Ecoli thymidine phoshorylase encapsulated within autologous erythrocytes

SUMMARY:
The purpose of this study is to determine the safety, tolerability, action and effectiveness of repeated doses of Erythrocyte Encapsulated Thymidine Phosphorylase (EE-TP) for the treatment of patients with Mitochondrial Neurogastrointestinal Encephalomyopathy (MNGIE).

MNGIE is a rare inherited disease that mainly affects the digestive and nervous system and is caused by a defect in the function of an enzyme called thymidine phosphorylase. This loss of function causes certain molecules (thymidine and deoxyuridine) to accumulate in cells which leads to toxic damage to these cells. The disease can be confirmed by detecting variations (mutations) in the thymidine phosphorylase gene (TYMP). Currently there are no specific treatments for patients with MNGIE, whose effectiveness has been shown through clinical trials. The potential treatment for MNGIE offered in this trial is an enzyme replacement therapy, i.e. replacing functional thymidine phosphorylase. This treatment uses the patients own red blood cells in which thymidine phosphorylase is encapsulated to produce EE-TP (the study drug). EE-TP is created using a machine named a Red Cell Loader (RCL) and is then administered back to the patient.

DETAILED DESCRIPTION:
This is a multi centre, multiple dose, open label study to investigate the safety, tolerability, pharmacodynamics and efficacy of EE-TP in patients with MNGIE. The study will be conducted in an open label manner with all patients receiving EE-TP.

The study will enrol 12 adult treatment naïve patients with MNGIE, aged 18 years or older at Screening. With Independent Data Monitoring Committee (IDMC) approval, a further four juvenile patients (aged 16-17) will be recruited after at least 24 patient-months exposure to treatment. With IDMC approval, a further four juvenile patients (aged 12-15) will be recruited after at least 24 patient-months exposure to treatment in the 16-17 year old patient group.

Screening failures and patients withdrawing from the study may be substituted with IDMC approval. Patients who have previously received EE-TP on a 'compassionate use' basis may be included in the study, if they meet eligibility criteria; these patients will be additional and will not be included in the sample size of 12.

The total sample size of 12 adult treatment naïve patients is not based on a formal statistical assessment, but is dictated by practical considerations mainly due to the rarity of the condition.

All patients will be administered EE-TP by intravenous (IV) infusion. There are 3 planned dose levels:

* Dose Level 1 (low dose): ~58 -65 x10^10 erythrocytes encapsulating 30 to 49 U TP/10^10 erythrocytes
* Dose Level 2 (mid dose): ~58 -65 x10^10 erythrocytes encapsulating 50 to 69 U TP/10^10 erythrocytes
* Dose Level 3 (high dose): ~58 -65 x10^10 erythrocytes encapsulating 70 to 90 U TP/10^10 erythrocytes

All patients will receive infusions at Dose Level 1 (low dose) for the first 2 treatment cycles. If metabolic correction is not achieved, the subsequent 2 treatment cycles will be infusions at Dose Level 2 (mid dose). If metabolic correction is still not achieved, treatment will advance to Dose Level 3 (high dose) for subsequent treatment cycles. If, at any time during this progression, metabolic correction is achieved, the patient will continue at the Dose Level in which metabolic correction has been achieved and there will be no further dose escalation.

Metabolic correction is defined as plasma thymidine <3 µmol/L and deoxyuridine <5 µmol/L (i.e., below the diagnostic levels for MNGIE).

The doses listed represent the planned doses; the starting dose will be Dose Level 1. It is anticipated that the highest dose will not exceed Dose Level 3; however, if metabolic correction is not achieved for an individual patient at this dose level, other modifications of dosing, such as increasing the number of erythrocytes administered in each infusion can be made.

Patients will be administered EE-TP every 3 weeks until the dose level achieving metabolic correction is identified. From Day 78 (or once metabolic correction has been achieved), it is planned that patients will receive EE-TP every 2 to 4 weeks until the end of the study. The interval between doses will not be shorter than 2 weeks ± 2 days. Dose selection will be flexible; continued pharmacodynamic assessment will enable dose optimization and further inform dose response models and establish the therapeutic window for the treatment.

Single doses of EE-TP will be administered on Day 0 then every 3 weeks until metabolic correction is achieved. The starting dose will be Dose Level 1, with potential subsequent dose levels of Dose Level 2 and Dose Level 3 dependent on whether metabolic correction is achieved or not. All doses will be administered IV.

From Day 78 (or once metabolic correction has been achieved), it is planned that patients will receive EE-TP every 2 to 4 weeks until the end of the study. Dose frequency may be reduced (e.g., from every 2 weeks to every 3 to 4 weeks) for individual patients based on ongoing review of emerging safety, tolerability, efficacy, and pharmacodynamic data. The interval between doses will not be shorter than 2 weeks ±2 days.

The dose level from day 78 onward will remain at the dose that achieved metabolic correction during the initial treatment phase (pre-day 78). In the advent of an increase in plasma metabolite levels (i.e. loss of metabolic correction), the frequency of dosing and/or dose level will be reviewed and adjusted accordingly.

Infusions with EE-TP will occur once every 2 to 4 weeks for 24 months.

Planned Enrolment/Screening (Run in) Duration: approximately 28 days (Days 120 to Day 92). Run-in period of 90 days (Days -91 to 0) for repeated evaluations of a number of assessments. Follow up, 90 days post dose. Planned Study Conduct Duration: approximately 31 months including screening, run-in period and post dose follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be male or female, of any race, aged 18 years or older at Screening.

   • Having IDMC reviewed the benefit risk profile and recommended progression to juvenile cohorts the age range will be extended to include patients:
   * aged 16 years or older after at least 24 patient months of exposure in patients aged 18 years or over.
   * aged 12 years or older after at least 24 patient months of exposure in patients aged <18 years at the time of enrolment.
2. Patients must be diagnosed with MNGIE by demonstrating all of the following:

   * <18% normal thymidine phosphorylase activity in the buffy coat;
   * >3 μmol/L plasma thymidine;
   * >5 μmol/L plasma deoxyuridine;
   * Confirmation of the presence of a pathogenic mutation in TYMP by sequencing.
3. Patients must be able to undergo study procedures.
4. Patients must agree to either remain completely true abstinent or to use 2 effective contraceptive methods from Screening until completion of the Follow up Visit
5. Patients must be willing to sign and date the written informed consent form after the benefits and risks of taking part in this study have been explained to them, and to comply with the study restrictions.

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible to participate in the study:

1. Patients who have received a successful liver or bone marrow transplant.
2. Patients suitable for allogeneic haematopoietic stem cell transplantation (AHSCT).
3. Patients with a matched AHSCT donor.
4. Patients with a known history of human immunodeficiency virus, hepatitis B infection, or an active hepatitis C infection.
5. Patients who are severely disabled (e.g., patient bed bound, incontinent, and unable to carry out any daily activities), or with a life expectancy of less than 12 months at Screening, based on the Investigator's judgment.
6. Female patients who are:

   * pregnant, planning a pregnancy, or are unwilling to use contraception
   * breastfeeding or lactating.
7. Patients who have donated blood in the 90 days prior to Screening.
8. Patients with a confirmed red blood cell count of <3.0 × 10^9 per mL.
9. Patients who have a significant history of alcoholism or drug/chemical abuse within 1 year prior to Screening, as determined by the Investigator.
10. Patients who have an abnormality in heart rate, blood pressure, or body temperature at Screening that, in the opinion of the Investigator, increases the risk of participating in the study.
11. Patients who have an abnormality in the 12 lead electrocardiogram (ECG) at Screening that, in the opinion of the Investigator, increases the risk of participating in the study.
12. Patients who have, or have a history of, any clinically significant neurological, GI, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological, or other major disorder (except for MNGIE, or disorders associated with MNGIE that, in the Investigator's opinion, do not constitute a risk when taking study drug and would not interfere with the study objectives) as determined by the Investigator.
13. Patients with any current malignancy, or a history of malignancy within 5 years prior to Screening, with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
14. Patients who are currently enrolled in, or are planning to participate in, or discontinued within the last 30 days from a clinical study involving an investigational medicinal product or concurrently enrolled in medical research judged not to be scientifically or medically compatible with EE-TP.
15. Patients with any medical condition, which in the opinion of the Investigator, would make the patient unsuitable for enrolment or could interfere with the patient's participation in, or completion of, the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The safety of EE-TP as measured by the incidence, frequency, and severity of treatment emergent adverse events | Day -120 to Follow-up visit (90 days post-final dose) at 31 months
  Incidence, frequency, and severity of adverse events will be summarised by dose level, maximum severity, and , Medical Dictionary for Regulatory Activities system organ class, and preferred term. The intensity/severity will be graded by Common terminology criteria for adverse events (CTCAE) criteria, including relation to treatment (IMP and/or infusion).
The safety of EE-TP as measured by the incidence of laboratory abnormalities, based on haematology, serum biochemistry, and urinalysis test | Day -120 to Follow-up visit (90 days post-final dose) at 31 months
  Incidence of laboratory abnormalities outside the clinical reference ranges based on haematology, serum biochemistry, and urinalysis test
The safety of EE-TP as measured by the vital sign measurements systolic and diastolic blood pressure | Day -120 to Follow-up visit (90 days post-final dose) at 31 months
  Systolic and diastolic blood pressure measured in units of millimeters of mercury (mmHg) will be recorded. Measurements outside the clinical reference ranges will be summarised by dose level, together with changes from baseline.
The safety of EE-TP as measured by the vital sign measurement heart rate | Day -120 to Follow-up visit (90 days post-final dose) at 31 months
  Heart rate measured as beats per minute (BPM) will be recorded. Measurements outside the clinical reference ranges will be summarised by dose level, together with changes from baseline.
The safety of EE-TP as measured by the vital sign measurement respiratory rate | Day -120 to Follow-up visit (90 days post-final dose) at 31 months
  Respiratory rate measured as number of breaths taken per minute will be recorded. Measurements outside the clinical reference ranges will be summarised by dose level, together with changes from baseline.
The safety of EE-TP as measured by the vital sign measurement body temperature | Day -120 to Follow-up visit (90 days post-final dose) at 31 months
  Body temperature measured in degrees Celsius will be recorded. Measurements outside the clinical reference ranges will be summarised by dose level, together with changes from baseline.
The safety of EE-TP as measured by 12 lead ECG parameters | Day -120 to Follow-up visit (90 days post-final dose) at 31 months
  12 lead ECG parameter data (QTc, QTcB, QTcF, the PR and QT intervals, QRS duration, and heart rate) outside the clinical reference ranges will be summarised by dose level.
The safety of EE-TP as measured by the use of concomitant medication(s) | Day -120 to Follow-up visit (90 days post-final dose) at 31 months
  The use of concomitant medication(s) will be listed
The assessment of pharmacodynamic effects of EE-TP by the measurement of plasma thymidine and deoxyuridine concentrations | Plasma and urine metabolites: Day -120 to Follow-up visit at 31 months
  Changes from baseline in plasma concentrations of thymidine and deoxyuridine will be calculated using Day 0 or Day 1 as the baseline.
The assessment of pharmacodynamic effects of EE-TP by the measurement of urine thymidine and deoxyuridine concentrations | Plasma and urine metabolites: Day -120 to Follow-up visit at 31 months; antibodies Day -1 to follow-up visit at 31 months
  Changes from baseline in urine concentrations of thymidine and deoxyuridine will be calculated using Day 0 or Day 1 as the baseline.
The efficacy of EE-TP as measured by change in body mass index (BMI) by recording weight and height | Study day -120 to end of study treatment at 24 months
  Body weight in Kilograms (Kg), in underclothes will be recorded at the same time of day using calibrated equipment.
  In patients aged 18 years or older, height in meters (m) will only be measured during Run-in and at Follow-up.
  In juvenile patients, height will be measured at all time-points with weight from Screening until Day 77, and every 3 months once metabolic correction has been achieved.
  BMI will be calculated by an individual's body mass divided by the square of his/her height [kg/m2]. Absolute and changes from baseline in BMI will be plotted against plasma and urine concentrations of thymidine and deoxyuridine.

SECONDARY OUTCOMES:
To assess the immunogenicity of EE-TP by monitoring the development of anti-thymidine phosphorylase antibodies | Baseline (Day -91 to Day 0) to end of study treatment at 24 months
  The presence of specific anti-thymidine phosphorylase antibodies will be recorded
To assess changes in clinical assessments as measured by total parenteral nutrition use | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  Total parenteral nutrition use will be recorded.
To assess changes in clinical assessments as measured by Handgrip strength using handgrip dynamometry | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  Handgrip strength measured using hand grip dynamometry (for assessment of distal muscle weakness) will be employed according to the Southampton protocol for adult grip strength.
To assess changes in clinical assessments as measured by Disability measured using the Rasch built Overall Disability Scale (RODS) | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  Multifocal motor neuropathy measured using the Rasch built Overall Disability Scale (RODS). This is a structured questionnaire containing 24 items that assesses activity and social participation limitation and graded as follows:
  0 = impossible to perform
  1. = performed with difficulty
  2. = easily performed
  A low score = worsening disability
To assess changes in clinical assessments as measured by ambulatory function measured using the timed 10 metre walk test | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  The 10 metre walk test measure will be used to assess walking speed in metres per second over a short distance. Patients will walk without assistance for 10 metres (32.8 feet) and the time will be measured from 6 metres (19.7 feet; to allow for acceleration and deceleration). The 'start time' will be when the toes of the leading foot cross the 2 meter mark. The 'stop time' will be when the toes of the leading foot cross the 8 meter mark.
  The 10 meter walk test will be performed at the preferred walking speed or at the fastest speed and performed 3 times, with the average calculated.
To assess changes in clinical assessments as measured by Clinical Global Impression - Improvement Scale (CGI I) | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  Quality of life measured using the Clinical Global Impression - Improvement Scale (CGI I)
  The CGI-I will provide a global measurement of the severity of a patient's clinical condition and improvement or worsening during the clinical study. The Investigator will assess the patient's condition relative to a 7 point scale ranging from 1 to 7:
  1. = very much improved
  2. = much improved
  3. = minimally improved
  4. = no change
  5. = minimally worse
  6. = much worse
  7. = very much worse Each component of the CGI is rated separately; the instrument does not yield a global score.
To assess changes in clinical assessments as measured by Quality of life measured using EuroQol 5-dimensions | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  EuroQol 5D consisting of 5 dimensions measuring generic health status; mobility, self care, usual activities, pain and discomfort, and anxiety and depression are all used to measure Quality of Life. Each dimensions consists of 5 levels of grading:
  no problem slight problem moderate problem severe problem extreme problem. When completing the questionnaire, patients will be required to assign the correct grade for the questions present.
To assess changes in clinical assessments as measured by gastrointestinal Symptoms symptoms using the Patient Reported Outcomes Measurement Information System (PROMIS) short form scales | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  Gastrointestinal (GI) symptoms will be assessed using the PROMIS short form scales:
  GI belly pain GI diarrhoea GI disrupted swallowing GI gas and bloating GI gastroesophageal reflux GI nausea and vomiting For the assessment of 'bothersome' and 'interference' of GI symptoms, a 5 point categorical response scale ranging from 'not at all' to 'very much' will be employed. For assessment of 'frequency,' a 5 level frequency scale will be employed. For assessment of 'bowel controllability,' a 5 level capability scale ranging from 'without any difficulty' to 'unable to control' will be employed, and for other items, unique response sets that optimally suit the concept of interest will be used as necessary.
  A score of 50 represents the average for a healthy state; a higher score represents a worse outcome and a lower score better than average.
To assess changes in clinical assessments as measured by Patient Global Impression of Change (PGIC). | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  Aspects of the patient's health will be measured using the PGIC which uses a 7-point scale to assesses if there has been an improvement or decline in clinical status:
  1. = very much improved
  2. = much improved
  3. = minimally improved
  4. = no change
  5. = minimally worse
  6. = much worse
  7. = very much worse PGIC assesses change in the severity of a patient's illness over a particular time interval
To assess changes in clinical assessments as measured by reflex responses using neurological examination tests | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  The reflex responses in:
  jaw jerk trigeminal nerve biceps brachioradialis triceps finger jerk knee jerk ankle jerk will be assessed according to the following 5 point scale: Grade 0 = no response; always abnormal, Grade 1+ = a slight but definitely present response; may or may not be normal, Grade 2+ = a brisk response; normal, Grade 3+ = a very brisk response; may or may not be normal, Grade 4+ = a tap elicits a repeating reflex (clonus); always abnormal.
To assess changes in clinical assessments as measured by muscle strength using the MRC scale | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  Muscle strength will be assessed according to the MRC scale in shoulder abduction, elbow flexion, wrist extension, first finger abduction, hip flexion, knee extension, and ankle dorsiflexion (MRC-sum 7 score) Grade 0 = no contraction Grade 1 = flicker or trace of contraction Grade 2 = active movement, with gravity eliminated Grade 3 = active movement against gravity Grade 4 = active movement against gravity and resistance Grade 5 = normal power
  Scores range from 0 (total paralysis) to 80 (normal strength).
To assess changes in clinical assessments as measured by sensory impairment scoring | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  Sensory impairment will be assessed using light touch, joint position sense, vibration sense, and pinprick using the following 3 point scale:
  Grade 0 = absent Grade 1 = impaired Grade 2 = normal
  A low score represents sensory disability.
To assess changes in clinical assessments as measured by improvement of the most disabling symptom for each patient using the visual analogue scale (VAS) | Change from baseline (Day -91 to Day 0) to end of study treatment at 24 months
  Improvement of the most disabling symptom for each patient will be assessed using the VAS which consists of a 20 cm vertical scale from 0 to 100, with the top end of the scale indicating the best health and the bottom end of the scale indicating the worst health. Patients will be required to identify a point on the scale to provide details of their health status.

OTHER OUTCOMES:
Exploratory Objective: to assess the effects of EE-TP on serum and plasma biomarkers of mitochondrial condition | Days 0, 1, 7, 14, 21, 28, 35, 42, 43, 49, 56, 63, 64, 70, and 77, and at each clinic visit from Day 78 until the end of the study
  Serum and plasma concentrations of biomarkers related to mitochondrial health such as fibroblast growth factor 21, growth differentiation factor 15, and other markers of mitochondrial condition will be measured longitudinally to determine any changes in response to therapy.
Exploratory Objective:to assess the effects of EE-TP on MRI brain | Change from baseline (Day -91 to Day 0) to 12 and 24 months
  MRI assessment of the head will be performed by qualified personnel
Exploratory Objective:to assess the effects of EE-TP on abdominal ultrasound | Change from baseline (Day -91 to Day 0) to 12 and 24 months
  Abdominal ultrasound examination will be performed by qualified personnel r
Exploratory Objective:to assess the effects of EE-TP on nerve conduction and Electromyography | Change from baseline (Day -91 to Day 0) to 12 and 24 months
  Nerve conduction studies will assess motor conduction velocity and sensory nerve conduction velocity. These tests will be used to diagnose MNGIE associated neuropathy. A needle electromyography will test the electrical activity of muscles, and help identify associated myopathy.
Exploratory Objective:to assess the effects of EE-TP on neuro ophthalmological assessments | Change from baseline (Day -91 to Day 0) to 12 and 24 months
  Neuro ophthalmological assessments (Hess chart and ptosis measurements as a minimum) will be performed to evaluate the relationship between the eye and the brain, and will include testing of visual acuity and colour vision, evaluation of eye movements and ocular alignment, and visual field testing.

CONTACTS AND LOCATIONS:
Overall Officials: Niranjanan Nirmalananthan, MBBS, Principal Investigator — St George's Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Moran NF, Bain MD, Muqit MM, Bax BE. Carrier erythrocyte entrapped thymidine phosphorylase therapy for MNGIE. Neurology. 2008 Aug 26;71(9):686-8. doi: 10.1212/01.wnl.0000324602.97205.ab. No abstract available. PMID 18725595
- [Result] Bax BE, Bain MD, Scarpelli M, Filosto M, Tonin P, Moran N. Clinical and biochemical improvements in a patient with MNGIE following enzyme replacement. Neurology. 2013 Oct 1;81(14):1269-71. doi: 10.1212/WNL.0b013e3182a6cb4b. Epub 2013 Aug 21. PMID 23966250
- [Result] Bourgeaux V, Lanao JM, Bax BE, Godfrin Y. Drug-loaded erythrocytes: on the road toward marketing approval. Drug Des Devel Ther. 2016 Feb 11;10:665-76. doi: 10.2147/DDDT.S96470. eCollection 2016. PMID 26929599
- [Result] Pacitti D, Levene M, Garone C, Nirmalananthan N, Bax BE. Mitochondrial Neurogastrointestinal Encephalomyopathy: Into the Fourth Decade, What We Have Learned So Far. Front Genet. 2018 Dec 21;9:669. doi: 10.3389/fgene.2018.00669. eCollection 2018. PMID 30627136